CLINICAL TRIAL: NCT01845753
Title: Molecular Screening for Lynch Syndrome in Denmark
Status: Completed | Type: Observational
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MS-LS-DK-02
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Colorectal Cancer; Lynch Syndrome; HNPCC
MeSH Terms: conditions — Colorectal Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All colorectal cancer patients
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observation

SUMMARY:
A clinically applicably strategy for molecular screening for Lynch Syndrome is being implemented in Denmark.

Based on sequential analysis with immunohistochemistry and methylation analysis, patients with possible hereditary colorectal cancer are identified. These patients are offered genetic risk assessment and counselling.

The study hypothesis is that molecular screening will identify more patients with Lynch Syndrome than the family history alone.

Prospective data collection is performed using established clinical databases.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of colorectal adenocarcinoma
* Diagnosed at one of the departments of pathology in Denmark

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All colorectal cancer patients in Denmark
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of Lynch Syndrome in a population of primary colorectal cancer | 1 year

CONTACTS AND LOCATIONS:
Locations (11):
- Denmark (11):
  - Department of Pathology, Aalborg
  - Department of Clinical Genetics, Aarhus
  - Department of Pathology, Aarhus
  - Department of Pathology, Esbjerg
  - Department of Pathology, Hjørring
  - Department of Clinical Genetics, Odense
  - Department of Pathology, Odense
  - Department of Pathology, Sønderborg
  - Vejle Hospital, Vejle
  - Department of Clinical Genetics, Vejle
  - Department of Pathology, Vejle